CLINICAL TRIAL: NCT04316039
Title: Radiotherapy Versus Radiotherapy Combined With Temozolomide in High-risk Low-grade Gliomas After Surgery
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Xingchen Peng, PhD, Associate Professor, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ChiCTR1800015199
Record Dates: First submitted 2020-03-17; First posted 2020-03-20 (Actual); Last update posted 2020-03-20 (Actual); Status verified 2020-03

CONDITIONS: Low-grade Glioma
Keywords: low-grade glioma; High-risk; Radiotherapy; Temozolomide
MeSH Terms: interventions — Temozolomide; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RT+TMZ (Experimental)
  Interventions: Drug: Temozolomide; Radiation: intensity modulated radiation therapy
- RT (Active Comparator)
  Interventions: Radiation: intensity modulated radiation therapy

INTERVENTIONS:
Drug: Temozolomide — Concurrent chemotherapy is to receive oral temozolomide, 75 mg/m2 per day, during radiation therapy. Adjuvant chemotherapy will be treated with six cycles of temozolomide, 150 to 200 mg/m2 per day for five consecutive days, repeated every 4 weeks. There is a 28-day break during radiotherapy and adjuvant temozolomide.
  Arms: RT+TMZ
Radiation: intensity modulated radiation therapy — The radiation dose is 50-54 Gy given in 25-30 fractions (1.8-2.0 Gy once daily, 5 days per week).

SUMMARY:
It has been reported that radiation therapy followed by PCV chemotherapy (procarbazine, lomustine and vincristine) could improve progression-free survival (PFS) and overall survival (OS) in patients with high-risk WHO grade 2 gliomas after surgery. However, procarbazine is not available in China. In clinical practice, Chinese doctors often use radiotherapy combined with temozolomide to treat these patients, though large-scale prospective studies are lacking. This trial aims to confirm whether RT combined with temozolomide can improve PFS and OS in patients with high-risk low-grade gliomas.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed supratentorial WHO grade II gliomas;
2. Aged 18 to 39 years without total resection, or aged 40 to 70 years with any extent of resection or biopsy;
3. Karnofsky performance score (KPS) ≥ 60;
4. No more than moderate neurologic symptoms and signs;
5. The interval between surgery and randomization is less than 12 weeks;
6. Have signed the consent form. -

Exclusion Criteria:

1. WHO grade I gliomas or high-grade gliomas according to WHO's grading system;
2. Have received prior radiation therapy to the head and neck region;
3. Have received prior chemotherapy;
4. Synchronous multiple primary malignant tumor excluding carcinoma of the cervix in situ or nonmelanomatous skin cancer;
5. Prior malignancy's disease-free survival less than 5 years;
6. Have active infection;
7. Patients are pregnant or breast-feeding. -

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2018-04-10 (Actual); Primary Completion 2023-04-10 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | up to 120 months
  Our primary outcome is progression-free survival which is calculated from the date of randomization to the date of first reported disease progression or the date of death.

CONTACTS AND LOCATIONS:
Overall Officials: Xingchen Peng, Ph.D, Principal Investigator — West China Hospital
Locations (1):
- Xingchen Peng, Chengdu, Sichuan, China